CLINICAL TRIAL: NCT02842268
Title: Evaluation of Sunscreen During Exercise Under Conditions of Profuse Sweating
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Bayer (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Other
Other Study IDs: 18818
Record Dates: First submitted 2016-06-20; First posted 2016-07-22 (Estimated); Last update posted 2018-12-13 (Actual); Status verified 2018-12

CONDITIONS: Sunscreening Agent

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- BAY987517 (Experimental): Subject will self-apply the test sunscreen formula to his/her face with the goal of applying 0.65 to 0.85 grams.Subject should sweat profusely.
  Interventions: Drug: BAY987517

INTERVENTIONS:
Drug: BAY987517 — Test product dried for at least 15 minutes.Subjects to ride for 30 minutes on a stationary bicycle.(Formulation Number :Y73-161)

SUMMARY:
To visually evaluate the retention of coverage of the Test Product(s) (TP) on the face after exercise compared to the full coverage observed prior to exercise.

ELIGIBILITY:
Inclusion Criteria:

* Subjects may be male or female, of an age of 18-55 years inclusive.
* Subjects must be capable of understanding and providing written informed consent.
* Subjects must sign a written confidentiality agreement including a photography release form.
* Subjects must be in good general health as judged by a specified licensed physician, who will indicate their suitability to participate in this study.
* Female subjects must be willing to take a rapid screen pregnancy test prior to each exercise session.
* Subjects must be willing to follow study instructions as set forth in the protocol.
* Subjects must not have facial piercing(s).
* Subjects must be Fitzpatrick Skin Type I, II, or III.

Exclusion Criteria:

* Subjects must not have received or used an Investigational New Drug within the last 30 days.
* Subjects must not have been active participants in another clinical or subjective TP performance study within the last 30 days unless authorized by this Sponsor.
* Subjects must not have a known physical or medical condition that would preclude vigorous exercise
* Subjects must not have a five-minute resting pulse rate greater than 80 bpm.
* Subjects must not take any chronic medication other than vitamins, hormone replacement therapy, low-dose aspirin, or oral contraceptives.
* Subjects must not have applied prescription or over-the-counter medicines to their face at least 96 hours prior to exercise session
* Subjects must not have a known allergy or sensitivity to sunscreen products or Cetaphil cleanser.
* Female subjects must not be pregnant (self-reported) or test positive using an on-site pregnancy test.
* Female subjects must not be nursing a child.
* Subjects must not have smoked cigarettes, pipes, or cigars in the last 60 days.
* Subjects who in the judgment of the Investigator have any condition that would make study participation inappropriate.
* Subjects must not be a member or relative of the clinical trial staff or the Sponsor directly involved in the study.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 15 (Actual)
Dates: Start 2016-06-17 (Actual); Primary Completion 2016-06-22 (Actual); Study Completion 2016-06-22 (Actual)

PRIMARY OUTCOMES:
Change of face coverage post exercise compared to the full coverage observed prior to exercise (in percent). | At baseline and post exercise (30 minutes)
  Done with a Skin Scanner( before and after each exercise session) using the 11-point scale

SECONDARY OUTCOMES:
Eye Stinging on grading scale | Up to 30 mins
  On scale:0 = None,1 = Slight,2 = Mild,3 = Moderate, 4 = Severe

CONTACTS AND LOCATIONS:
Overall Officials: Bayer Study Director, Study Director — Bayer
Locations (1):
- St. Petersburg, Florida, United States